CLINICAL TRIAL: NCT03191357
Title: Evaluation of Military Service and Family Members for Post Concussive and Posttraumatic Stress Symptoms
Acronym: MRP
Status: Completed | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MED-83-2622
Record Dates: First submitted 2017-06-12; First posted 2017-06-19 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2017-06

CONDITIONS: TBI (Traumatic Brain Injury)
Keywords: traumatic brain injury,posttraumatic stress,service member
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — During this study, no more than 40 mL or one ounce, of blood will be drawn. Participants may decline the blood draw and still participate in other study procedures. A phlebotomist, research nurse, or trained and credentialed study team member will draw samples. The samples sent directly to the CNRM Biospecimen Repository. WRNMMC samples will be transported by Runners Courier services. The FBCH samples will be packaged and shipped overnight FedEx directly to the Biospecimen Repository.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- TBI/no PH: Active and reserve component SMs along with others who are eligible for care in the DoD healthcare system, who have experienced traumatic brain injury (TBI) without psychological health (PH) concerns.
  no intervention/Observational
  Interventions: Other: n/a observational
- TBI with PH: Active and reserve component SMs along with others who are eligible for care in the DoD healthcare system, who have experienced traumatic brain injury (TBI) and also have psychological health (PH) concerns.
  no intervention/Observational
  Interventions: Other: n/a observational
- PH only: Active and reserve component SMs along with others who are eligible for care in the DoD healthcare system, who have experience psychological health (PH) concerns.
  no intervention/Observational
  Interventions: Other: n/a observational
- Controls: Control participants may include (i) those with exposure to primary blast without the development of TBI, (ii) those with physical injuries without experiencing head injury, and (iii) healthy participants (non-injured, non-TBI, non-PH).
  no intervention/Observational
  Interventions: Other: n/a observational

INTERVENTIONS:
Other: n/a observational — Observational study

SUMMARY:
This protocol is designed to facilitate the recruitment, screening and registry of Military Service Members (SMs) and individuals eligible for care in the Department of Defense (DoD) healthcare system. This protocol will serve as an entry point for SMs, retirees and other beneficiaries, to facilitate their participation in Center for Neuroscience and Regenerative Medicine (CNRM)-sponsored clinical research studies at participating CNRM sites. Specifically, this protocol will be comprised of an initial evaluation of participants, to include questionnaires, a blood draw, and neuroimaging. This evaluation will enable investigators to direct participants to CNRM-sponsored natural history, observational, or interventional protocols that are most relevant to the individual interests and needs of each participant. Other approved CNRM protocols may continue to recruit participants directly into their respective studies, and may refer participants to this study.

The objective of this protocol is to develop a broad-spectrum military subject recruitment database that will collect and store preliminary data on research participants who are interested in and potentially eligible for current and future CNRM sponsored studies. The effectiveness of the recruitment methods utilized in this protocol will be evaluated to determine the most successful outreach approaches and recruitment tools for the enrollment of participants, including both active and reserve component SMs along with others who are eligible for care in the DoD healthcare system, who have experienced traumatic brain injury (TBI), psychological health (PH) concerns, or are interested in participating in studies as controls. Control participants may include (i) those with exposure to primary blast without the development of TBI, (ii) those with physical injuries without experiencing head injury, and (iii) healthy participants (non-injured, non-TBI, non-PH).

DETAILED DESCRIPTION:
This protocol is designed to facilitate the recruitment, screening and registry of Military Service Members (SMs) and individuals eligible for care in the Department of Defense (DoD) healthcare system. This protocol will serve as an entry point for SMs, retirees and other beneficiaries, to facilitate their participation in Center for Neuroscience and Regenerative Medicine (CNRM)-sponsored clinical research studies at participating CNRM sites. Specifically, this protocol will be comprised of an initial evaluation of participants, to include questionnaires, a blood draw, and neuroimaging. This evaluation will enable investigators to direct participants to CNRM-sponsored natural history, observational, or interventional protocols that are most relevant to the individual interests and needs of each participant. Other approved CNRM protocols may continue to recruit participants directly into their respective studies, and may refer participants to this study.

The objective of this protocol is to develop a broad-spectrum military subject recruitment database that will collect and store preliminary data on research participants who are interested in and potentially eligible for current and future CNRM sponsored studies. The effectiveness of the recruitment methods utilized in this protocol will be evaluated to determine the most successful outreach approaches and recruitment tools for the enrollment of participants, including both active and reserve component SMs along with others who are eligible for care in the DoD healthcare system, who have experienced traumatic brain injury (TBI), psychological health (PH) concerns, or are interested in participating in studies as controls. Control participants may include (i) those with exposure to primary blast without the development of TBI, (ii) those with physical injuries without experiencing head injury, and (iii) healthy participants (non-injured, non-TBI, non-PH).

This protocol will serve four purposes: (i) provide a centralized resource to identify and screen individuals in order to facilitate their participation in ongoing CNRM studies, (ii) for participants who provide informed consent to do so, to confidentially and securely collect, store, and disseminate to other CNRM investigators existing personally identifiable information (PII), existing protected health information (PHI) and data collected as part of research under this protocol, (iii) provide a mechanism for following and contacting subjects for participation in future CNRM studies, and (iv) assess the impact of TBI and PH issues upon structural and functional imaging measures to provide a more comprehensive overview of participants being referred to other CNRM studies.

Research Design:

This is an "umbrella" cohort study designed to facilitate recruitment of military SMs and others eligible for care in the DoD healthcare system in order to collect preliminary data pertaining TBI, postconcussive syndrome (PCS), posttraumatic stress (PTS), and/or other PH concerns, along with comparable data on relevant control groups. Important control comparisons are a) those with exposure to primary blast without the development of TBI, b) those with other types of physical injuries without head injury exposure, and c) healthy controls. These control comparisons are necessary to address pertinent research questions on PCS and PTS. Based on the information provided by each participant, as well as their preferences expressed during their initial contact with study staff, each may either be directly referred to appropriate CNRM protocols, informed that he/she is not eligible for any other actively enrolling CNRM studies at this time, or proceed with full participation in this enrollment protocol.

Methodology/Technical Approach:

Over a 5-year period, this protocol seeks to enroll up to 2000 male and female SMs as well as others who are also eligible for care in the DoD healthcare system with signs and symptoms of TBI, PCS, PTS or PTSD and/or other PH concerns, or relevant controls (up to 25%, or 100 per year, may have exposure to primary blast without known development of TBI, physical injuries without evidence of head injury, and healthy controls). Up to 400 subjects per year over the next five years will be enrolled through either the standard or the abbreviated pathway and will undergo study procedures at the participating sites: Fort Belvoir Community Hospital (FBCH), including the Intrepid Spirit One and Brain Assessment Research Laboratory (BARL); Uniformed Services University of the Health Science (USUHS), including the Clinical Research Unit, (CRU) Clinical Psychophysiology and Psychopharmacology Laboratory (CPPL); and Walter Reed National Military Medical Center (WRNMMC), including Defense and Veterans Brain Injury Center (DVBIC) and BARL. Participants may also be enrolled in the abbreviated pathway from the CNRM site at Twinbrook, although other study procedures will not occur there.

The study will be composed of two research pathways: (i) a standard pathway and (ii) an abbreviated pathway. Prior to enrollment, both pathways will pre-screen potential participants to assess eligibility for the current study and for the protocol WRNMMC 353853. Information on the prescreen form is collected to assist with scheduling study assessments such as patient interviews and placing orders for imaging and blood collection. Participants eligible for the WRNMMC 353853 will have the option to dual enroll into that study. Parenthetically, it should be noted that WRNMMC 353853 recruits inpatients from the Neurology and Neurosurgery Service, as well as the Neurology Clinic at WRNMMC; while the current study encompasses many of the same procedures as WRNMMC 353853, the intent of the current study is to recruit a much broader population, including healthy controls, those with primary psychological health concerns, and those with blast exposure who do not necessarily meet criteria for TBI. To facilitate accrual of our cohort, we will actively recruit from a much broader range of settings, including primary care, behavioral health, and orthopedics and rehabilitation clinics at WRNMMC, and a wide array of clinics and services at FBCH, in addition to using CNRM's social media and other web-based efforts. Applicable study procedures will depend on the pathway for enrollment, diagnostic certainty, and logistic considerations such as distance from participating sites, availability of scanners, and feasibility of transport.

Standard Pathway: Visit procedures for this pathway will be conducted at the participating sites (FBCH, USUHS, WRNMMC) and will consist of informed consent, collection of PII/PHI, generation of a Global Unique Identifier (GUID) as detailed below in section 6.3.4., structured data collection of medical history, combat-related as well as any civilian injury details, symptom inventory, blood collection and validated questionnaires to assess symptoms. Scale cards containing the potential responses for each of the questionnaires will be provided to participants for in-person interviews. The scales correlate to specific study data collection measures (questionnaires). The scale cards will allow the participant to view the answer choices for each measure while the study team member administers the questionnaires. The scale cards will ensure greater participant understanding during administration of the questionnaires. Additionally, this pathway will include collection of venous blood and a MRI of the brain for participants who consent to these elements. Visit procedures will also include a physical exam, neurocognitive assessments, and exit consultation. See section 6.3 Study Design for further detail.

Abbreviated Pathway: Visit procedures for this pathway will consist of informed consent, collection of PII/PHI, generation of a GUID as detailed below in section 6.3.4., an abbreviated questionnaire for structured collection of a medical history, injury details, and validated questionnaires assessing symptoms. Scale cards containing the potential responses for each of the questionnaires will be mailed to participants for telephonic interviews. The scales correlate to specific study data collection measures (questionnaires). The scale cards will allow the participant to view the answer choices for each measure while the study team member administers the questionnaires. The scale cards will ensure greater participant understanding during administration of the questionnaires. Potential research participants will be enrolled in this abbreviated pathway by participating in a (i) telephonic interview or (ii) an in-person interview at Twinbrook, participating sites, or at recruitment events, or through some combination of these approaches. See section 6.3 Study Design for further detail.

Objectives:

The primary objective of this protocol is to facilitate recruitment of SMs and those eligible for care in the DoD healthcare system to CNRM sponsored clinical research at participating CNRM sites.

Additional aims of the study are to:

* Use data collected through this protocol to improve recruitment methods
* Coordinate the enrollment of participants in CNRM studies with the greatest relevance and interest to them, maintain longitudinal contact, and offer those who are interested the opportunity to participate in subsequent CNRM studies after enrollment in this study
* Use data collected through the neurocognitive assessment (NIH Toolbox) to better direct referral to appropriate CNRM studies
* Establish and maintain study specific recruitment databases containing (i) identifiable data (PII and PHI) and (ii) coded research data
* Collect and provide blood and de-identified data to IRB-approved CNRM Biospecimen and Informatics Repositories for use in future research studies (storage procedures covered by USUHS IRB protocol "Biorepository and Informatics Warehousing", CNRM 004)
* Assessment of TBI and psychological stress impact on the brain via structural and functional imaging as well as diffusion tensor imaging
* Assess imaging and neurocognitive data for patterns that could distinguish those with ongoing symptoms vs. those who are more resilient after trauma

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age.
2. Active duty, retired military SM, TRICARE eligible reservist or National Guardsman, or a family member eligible for care in the DoD healthcare system.
3. Ability to provide self-consent
4. For TBI participants, must report having symptoms or diagnosis of a concussion, TBI with or without loss of consciousness, or PCS; the duration of time since the head injury will be documented, but there is no limitation on duration since some CNRM studies do not place a time limit. Medical documentation is preferred but not required
5. For participants with psychological health concerns, must report having current symptoms or may already have a diagnosis of PTSD, depression, or generalized anxiety disorder.
6. For injured participants without TBI, must be (i) exposed to primary blast or (ii) have other orthopedic and/or soft-tissue injury for which they sought care at a medical treatment facility within the past six months. Injury sustained can be combat or non-combat related.
7. For healthy controls, must be healthy with no prior diagnosis of TBI, concussion, PTSD, and/or other PH issues, and no history of exposure to blast.
8. Are willing to have their contact information and data shared and stored by the CNRM for referral to current and future CNRM studies.

Exclusion Criteria:

1. Individuals who are unable to provide their own informed consent for the study
2. Individuals who are unwilling or unable to cooperate with study procedures
3. Individuals with penetrating brain injury with residual shrapnel or other MRI-incompatible metal embedded in the brain or skull (excluded from MRI only, can still take part in study)
4. Individuals with contraindication to MRI scanning including certain metal implants or devices (excluded from MRI only, can still take part in study)
5. Those with conditions precluding entry or prolonged durations in the MRI scanners, e.g. morbid obesity, severe claustrophobia, etc., (excluded from MRI only, can still take part in study)
6. Pregnancy: urine pregnancy tests will be performed on all females prior to the conduct of MRI; if a positive pregnancy test is identified, MRI will not be performed, can still take part in study.
7. Individuals with self reported psychosis, schizophrenia, schizoaffective disorder, bipolar disorder, conversion disorder or personality disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participant population for the study includes all active duty, retired military SMs, TRICARE eligible reservists or National Guard, or interested family members who are at least 18 years and eligible for care in the DoD healthcare system; participants may be of any racial or ethnic origin, gender, or sexual orientation.
Sampling Method: Probability Sample
Enrollment: 424 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Broad-spectrum military subject recruitment database | five years
  Capture data for up to 2000 male and female service members, as well as others who are also eligible for care in the DoD healthcare system, with signs and symptoms of TBI , PCS, PTS or PTSD and/or other PH concerns, or relevant controls. Assessments and procedures include self-report questionnaires, brief physical exam, neuroimaging, neurocognitive assessment, and blood sample collection. Data collected will be stored and managed by the CNRM data repositories.

SECONDARY OUTCOMES:
Improvement of recruitment methods | five years
  *Use enrollment data including neuroimaging, biospecimen, neurocognitive and self-reports coupled with retention and attrition data collected through this protocol to improve recruitment methods.
Enrollment and referral | five years
  *Coordinate the enrollment of participants in CNRM studies with the greatest relevance and interest to them, maintain longitudinal contact, and offer those who are interested the opportunity to participate in subsequent CNRM studies after enrollment in this study
Recruitment databases | five years
  *Use data collected through the neurocognitive assessment (NIH Toolbox) to better direct referral to appropriate CNRM studies

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Roy, MD, MPH, Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Uniformed Services University of Health Sciences (USUHS), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Information to be shared via Fitbir